CLINICAL TRIAL: NCT00920595
Title: An Open-Label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CEP-9722 (a PARP-1 and PARP-2 Inhibitor) as Single-Agent Therapy and as Combination Therapy With Temozolomide in Patients With Advanced Solid Tumors
Brief Title: Study of CEP-9722 as Single-Agent Therapy and as Combination Therapy With Temozolomide in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C9722/1065/PK/FR-UK; EudraCT number: 2008-006858-18
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Solid Tumor
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — CEP-9722

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CEP-9722 alone and in combination therapy with temozolomide.
  Interventions: Drug: CEP-9722

INTERVENTIONS:
Drug: CEP-9722 — Starting dose of CEP-9722 is 150 mg/day (total dose). The study consists of a 14-day cycle of CEP-9722 alone, and at least one 28-day cycle of CEP-9722 plus temozolomide (150 mg/m2/day on Days 1-5). Patients who are receiving clinical benefit may receive subsequent cycles of study drug treatment.

SUMMARY:
An open-label study to evaluate the safety, pharmacokinetics, and pharmacodynamics of CEP-9722 as single-agent therapy and as combination therapy with temozolomide in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a histologically or cytologically confirmed malignant advanced solid tumor considered unresponsive or poorly responsive to accepted treatment modalities.
* The patient has adequate hematologic assessments and adequate renal and hepatic functions as specified in the study protocol.
* The patient has measurable or nonmeasurable disease documented with an appropriate method of evaluation according to disease characteristics.
* The patient has had no chemotherapy for at least 3 weeks and has resolution of prior sequelae. If the patient has had prior curative radiation or prior treatment with nitrosoureas, a minimum of 4 weeks and 6 weeks, respectively, must have elapsed before treatment with CEP-9722.
* The patient has had no immunotherapy, including monoclonal antibody therapy, for at least 4 weeks and no hormonotherapy for at least 1 week, with the exception of patients with prostate cancer, who may continue hormonal therapy.
* The patient has a European Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* The patient has a life expectancy of 12 weeks or more.
* Agreement by women of childbearing potential (not surgically sterile or 2 years postmenopausal) to use a medically accepted method of contraception and continue the use of this method for the duration of the study and for 90 days after participation in the study. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* Agreement by men not surgically sterile or who are capable of producing offspring to practice abstinence or use a barrier method of birth control, and continue use of this method for the duration of the study and for 6 months after participation in the study.

Exclusion Criteria:

* The patient has a primary brain tumor whose disease requires a systematic premedication with anticonvulsive agents.
* The patient has baseline cardiac abnormalities outside of the specified study parameters.
* The patient has clinically symptomatic recurrent/progressive brain metastases within 4 weeks (stable sequelae are acceptable).
* The patient has previous hypersensitivity reactions to 1 of the components of CEP-9722, temozolomide, or dacarbazine.
* The patient is a pregnant or breast-feeding woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The patient is participating in another interventional clinical study at the time of enrollment, has participated in another interventional clinical study within 4 weeks prior to enrollment, or the patient has previously been already enrolled in this study.
* The patient has an active gastroduodenal ulcer, uncontrolled high blood pressure, uncontrolled diabetes mellitus, or uncontrolled angina pectoris; has had a recent myocardial infarction; has had a cerebrovascular event within 6 months prior to study entry; or has pre-existing coagulopathy.
* The patient has a concomitant uncontrolled infection or severe systemic disease.
* The patient has a known nephropathy or hepatopathy.
* The patient is receiving concurrent treatment with an antineoplastic agent other than temozolomide.
* The patient has had previous treatment with another PARP inhibitor.
* The patient is unable to swallow capsules.
* The patient has taken any medications which are contraindicated as specified in the study protocol.
* The patient has any serious or uncontrolled nonmalignant medical disorder or psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) upon Dose Limiting Toxicities (DLT) data | Up to 42 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Days 1 and 5 of Cycle 1 and on Day 5 of Cycle 2
Pharmacodynamics assay | Days 1, 5, and 8 of both Cycle 1 and Cycle 2
Efficacy - will be assessed by the proportion of patients who achieve tumor response during the study | A 14-day cycle and at least one 28-day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon France
Locations (2):
- Cephalon Investigational Site, Nantes, France
- Cephalon Investigational Site, Newcastle upon Tyne, United Kingdom